CLINICAL TRIAL: NCT03376581
Title: The Utility of Platelet Rich Plasma in Hair Loss
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Natasha Mesinkovska, Principal Investigator, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20163239
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Prospective treatment (Experimental)
  Interventions: Procedure: Platelet rich plasma

INTERVENTIONS:
Procedure: Platelet rich plasma — Blood drawn from each participant will be spun down to separate platelets. Platelets will be injected into that patient's scalp.

SUMMARY:
Platelet rich plasma (PRP) is an autologous preparation of human plasma with high concentration of platelets. Platelets release numerous growth factors, which stimulate cell proliferation and differentiation.

The purpose of this research is to investigate the potential of PRP injection for treatment of hair loss. Clinical outcomes will be assessed by noninvasive techniques including dermoscopy, multiphoton microscopy, optical coherence tomography, optical Doppler tomography and multispectral imaging.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Ability to understand and carry out instructions
* Diagnosed with alopecia

Exclusion Criteria:

* Inability to understand and.or carry out instructions
* Pregnant women
* Use of any topical medication (such as minoxidil or any other solution for hair growth), oral medication (finasteride, dutasteride, or antiandrogens), laser therapy, or chemotherapy, within the preceding 4 weeks.
* Personal medical history of bleeding disorders
* Personal medical history of platelet dysfunction syndrome
* Anti-coagulation therapy or nonsteroidal anti-inflammatory drugs in the last 1 week.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Hair density to measure the efficacy of treatment | 6 months

SECONDARY OUTCOMES:
Hair count (number of hairs/0.65 cm2) | 6 months
Terminal hair density | 6 months
Anagen hair percentage | 6 months
Telogen hair percentage | 6 months
Anagen/telogen ratio | After 3 and 6 months
Changes in hair structure, diameter, and blood flow | 6 months
  As measured by optical coherence tomography

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine, Department of Dermatology, Dermatology Clinical Research Center, Hewitt Hall, Irvine, California, United States